CLINICAL TRIAL: NCT02615379
Title: A Prospective, Randomized, Parallel Pilot Study of Transdermal, Continuous Oxygen Therapy for Infection Prophylaxis in High- Risk Patients Undergoing Instrumented Fusion
Brief Title: Transdermal Continuous Oxygen Therapy for Infection Prophylaxis in High- Risk Patients Undergoing Instrumented Fusion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Neogenix, LLC dba Ogenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EPF-515
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Instrumented Spinal Fusion
Keywords: instrumented spinal fusion; infection; topical oxygen
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be given blinded data and pictures to enable unbiased assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transdermal Continuous Oxygen Therapy (Experimental): EPIFLO® working study unit, all day, every day for 2 weeks + standard wound care
  Interventions: Device: EPIFLO
- Standard of care (No Intervention): standard wound care for 2 weeks

INTERVENTIONS:
Device: EPIFLO — Transdermal continuous oxygen therapy is oxygen delivery to the wound site directly. Ogenix makes a small portable oxygen concentrator (Trade Name: EPIFLO) that makes continuous transdermal delivery of oxygen possible. It is a 3 ounce oxygen generator that continuously delivers 3 ml of pure oxygen to the wound site.
  Other Names: TCOT, Transdermal Continuous Oxygen Therapy
  Arms: Transdermal Continuous Oxygen Therapy

SUMMARY:
EPIFLO® unit along with standard wound care vs only standard wound care for Surgical site infections (SSI).

DETAILED DESCRIPTION:
Surgical site infections (SSI) after instrumented spinal fusions are not rare, and patients with SSI after instrumented spinal surgery often require repeat operations and prolonged intravenous antibiotic therapy. Wound hypoxia has been identified as a pathogenic mechanism behind wound infection and poor healing. Transdermal oxygen delivery (EPIFLO) has recently become a novel strategy to facilitate wound healing.

The study doctor will give an EPIFLO® unit along with standard wound care to some subjects in this study to see if it is safe and can help them. Another purpose of this study is to find out if using EPIFLO® is better than getting only standard wound care for Surgical site infections (SSI). The sponsor also wants to compare the cost of using the study device and standard wound care to the cost of standard wound care alone. The U.S. Food and Drug Administration (FDA) has approved EPIFLO® to treat skin ulcers (including diabetic skin ulcers), bedsores, amputations, skin grafts, burns, and frostbite.

ELIGIBILITY:
Inclusion Criteria:

* Elective spinal fusion - posterior cervical, posterior thoracic, or posterior lumbar instrumented spinal fusions
* Patient Age 18-80
* Patients must be considered high risk for infection, meeting one or more of the following criteria:

  * Anticipated Surgical duration ≥ 3 hours
  * Diabetes Mellitus type I or II
  * Anesthesiology ASA score of 3 or above
  * BMI ≥35
  * Patients with malnutrition as indicated by Pre-albumin value of <20
  * Chronic corticosteroid use
  * Smokers
  * Patients on immune modulators

Exclusion Criteria:

Major Study Exclusion Criteria include:

* Pregnancy
* Active infection at the time of surgery
* Persons with decubitus or diabetic ulcers
* Patients undergoing >5 level fusion (Level is defined as crossing a disk space; e.g.,an L3-5 fusion is a 2 level fusion)
* Disseminated Cancer Patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site infection | 3 months
  The primary objective of this study is to assess surgical site infection within 3 months of surgery for "high risk" patients undergoing posterior cervical, posterior thoracic, or posterior lumbar instrumented spinal fusions in patients receiving adjunct Transdermal Continuous Oxygen therapy vs. standard of care control. Surgical site infection will be clinically assessed by the PI according to CDC criteria. Independent blinded assessment by a clinician blinded to the allocation arm will also be obtained. The number of patients with infection (and the severity of infection) in the treated arm will be compared to the number in the control arm.

SECONDARY OUTCOMES:
Resource utilization | 3 months
  Resource utilization- the sum total of cost of treatments, hospital stays, bandages, nursing care and anything else related to treatment all measured in dollar amounts and then summed
Severity of infection | 3 months
  Severity of infection - Superficial or deep as per CDC classification as assessed by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Tomycz, M.D., Principal Investigator — Department of Neurosurgery
Locations (1):
- Department of Neurological Surgery Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided